CLINICAL TRIAL: NCT05084456
Title: Weekly Administration of (bi-)Daily Oral Docetaxel in Combination With Ritonavir in Patients With Normal or Impaired Liver Function
Brief Title: Oral Docetaxel in Patients With Normal or Impaired Liver Function
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending further development
Sponsor: Modra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N16DOL
Record Dates: First submitted 2019-03-25; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor, Adult; Impaired Liver Function
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: At least 6 evaluable patients will be included in every of the three groups: a) Controls (Child-Pugh class A with normal biochemical liver tests), b) Child-Pugh class A patients with impaired biochemical liver tests, c) Child-Pugh class B patients. Therefore a minimum of 18 evaluable patients will be included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): ModraDoc006/r will be administered in a continuous weekly dose of 30-20 mg without dose escalation. This is the established recommended phase II dose for patients with normal liver function based on previous phase I trials.
  Interventions: Drug: ModraDoc006/r
- Child-Pugh class A (Experimental): ModraDoc006/r administration will start treatment with a weekly BID dose of 20-10mg ModraDoc006 in combination with ritonavir. If toxicity is acceptable, after 4 weeks an intra-patient dose-escalation will be initiated, followed by the second dose escalation after another 4 weeks.
  Interventions: Drug: ModraDoc006/r
- Child-Pugh class B (Experimental): ModraDoc006/r administration will start treatment with a weekly QD dose of 20mg ModraDoc006 in combination with ritonavir. If toxicity is acceptable, after 4 weeks an intra-patient dose-escalation will be initiated, followed by the second dose escalation after another 4 weeks.
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — Treatment with weekly ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets in fed or fasting condition
  Other Names: Oral docetaxel formulation

SUMMARY:
This is an open label, single centre pharmacological and safety study to define the safety and pharmacokinetics of ModraDoc006/r in a weekly dosing schedule in patients with impaired liver function who might have benefit from a weekly docetaxel regime. The safety of ModraDoc006 in combination with ritonavir for the patients with mild and moderate impaired liver function will be evaluated with a dose escalation design.

DETAILED DESCRIPTION:
Oral administration of (anticancer) drugs has many advantages above intravenously administered compounds for patients. A major obstacle for development of an oral docetaxel formulation is the observed poor bioavailability of the drug after oral administration. This was efficiently improved in several pre-clinical and early clinical studies by co-administration of the CYP3A4 inhibitor ritonavir and by development of a new oral formulation of docetaxel (ModraDoc006).

Currently, treatment with ModraDoc006/r (i.e. oral docetaxel as tablets of 10 mg combined with a ritonavir dose of 100 mg) has been evaluated in several clinical trials at the NKI. In these trials, patients have been treated with ModraDoc006/r for a duration of up to 72 weeks.

Commonly observed toxicities of ModraDoc006/r in the phase I trials were nausea, vomiting, diarrhea and fatigue, mostly being of CTC (Common Toxicity Criteria) grade 1-2 severity and usually not interfering with the therapy. Frequently occurring toxicities of intravenously administered docetaxel, such as neutropenia, hypersensitivity reactions and peripheral polyneuropathy have rarely been observed with ModraDoc006/r.

The established recommended dose for further treatment with ModraDoc006/r is 30mg ModraDoc006 (combined with 100mg ritonavir) in the morning and 20 mg ModraDoc006 (combined with 100 mg ritonavir) in the afternoon, as a bidaily weekly schedule.

Impaired hepatic function The primary goal of this study is to explore the safety and pharmacokinetics of ModraDoc006/r in patients with mild or moderate liver impairment in order to be able to give appropriate and practical dose recommendations in daily clinical practice. According to the recommendations of the EMA and FDA guidelines, the Child-Pugh classification will be used in this study to define different classes of severity of liver impairment. However, patients with Child-Pugh class C score will not be included in the study, because of the expected poor performance status and survival and expected increased toxicity related to severely impaired organ function, for whom the use of ModraDoc006/r is considered contra-indicated.

Patients will receive oral docetaxel (as ModraDoc006 10 mg tablets) and ritonavir (100 mg tablet) once- or bi-daily, once a week in a fasted condition. After the end of the study period of twelve weeks patients will go off study and will immediately be offered the opportunity to embark on the roll over protocol N17DEX. This will ensure fully that the patient will receive ModraDoc006/r in the best interest without limitations.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of cancer
2. Patients who might benefit from a weekly (oral) docetaxel regime
3. One of the following options regarding liver impairment:

   * Normal liver function: Child-Pugh A classification and normal (<ULN) values of total bilirubin and ASAT/ALAT)
   * Presence of liver impairment according to the following characteristics:

     * Child-Pugh A and elevated (>ULN) values of total bilirubin and/or ASAT/ALAT (as described in table 3 or Appendix VI)
     * Child-Pugh B
4. Age ≥ 18 years;
5. Able and willing to give written informed consent;
6. WHO performance status of 0, 1 or 2;
7. Able and willing to undergo blood sampling for PK analysis;
8. Life expectancy > 3 months;
9. Minimal acceptable laboratory values defined as:

   1. Hb ≥ 6.0 mmol/L
   2. ANC of ≥ 1.5 x 109 /L
   3. Platelet count of ≥ 100 x 109 /L
   4. Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula);
10. Negative pregnancy test (urine/serum) for female patients with childbearing potential;
11. Able and willing to swallow oral medication

Exclusion Criteria:

1. Severe liver impairment classified as Child-Pugh C
2. Concomitant use of anticoagulant drugs that can or do alter the PT-INR
3. Other causes of elevated bilirubin than intrinsic liver impairment (as described in appendix VII)
4. Concomitant use of MDR and CYP3A modulating drugs such as Ca+-entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, quinine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications; other protease inhibitors, (non) nucleoside analoga, St. Johns wort or macrolide antibiotics.
5. Bowel obstructions or motility disorders or gastrectomy that may influence the absorption of drugs
6. Neurologic disease that may render a patient at increased risk for peripheral or central neurotoxicity
7. Patients with symptomatic brain metastases or with leptomeningeal metastases. Patients with brain metastases are allowed if they received adequate treatment, are asymptomatic in the absence of corticosteroid therapy and anticonvulsant therapy for at least 6 weeks. Radiotherapy for brain metastases must have been completed at least 4 weeks prior to start of study treatment. Brain metastases must be stable with verification by imaging (e.g. brain MRI or CT completed at screening).
8. Unresolved > grade 1 toxicities of previous systemic therapy, except for alopecia
9. Woman who are pregnant or breast feeding;
10. Unreliable contraceptive methods. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms)
11. Radio- or chemotherapy or any treatment with investigational drugs within the last 4 weeks prior to receiving the first dose of investigational treatment (palliative limited radiation for pain reduction is allowed);
12. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
13. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance;
14. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications;
15. Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The AUC of docetaxel (area under the curve) | Pharmacokinetic plasma sampling during 48 hours in Cycle 1 and Cycle 5 (each cycle is 7 days)
  The AUC of docetaxel given as bi-daily ModraDoc006 10 mg tablets in combination with ritonavir after administration in patients with normal and impaired liver function
The hematological and non-hematological toxicity profile of oral docetaxel in combination with ritonavir | Safety and tolerance will be evaluated during the complete study treatment untill 28 days after the last intake, using the CTCAEv4.03 grading system
  The number of CTCAE v.4.03 grade 3-4 toxicities during treatment with ModraDoc006/r

CONTACTS AND LOCATIONS:
Overall Officials: Serena Marchetti, MD/PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No